CLINICAL TRIAL: NCT01665599
Title: A Phase 3, Open-label, Non-randomized, Clinical Trial to Evaluate the Efficacy and Safety of FE 999303 (Testosterone Gel) in Adult Hypogonadal Males
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Testosterone Gel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000023
Record Dates: First submitted 2012-08-01; First posted 2012-08-15 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Adult Male Hypogonadism
MeSH Terms: conditions — Eunuchism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone gel (FE 999303) (Experimental): Subjects received a starting dose of 46 mg (two actuations) of testosterone gel (2%) daily in the morning. The dose was further titrated (increased or decreased - three actuations [69 mg] or single actuation [23 mg], respectively) based on serum testosterone concentrations.
  Testosterone gel was applied using an applicator, to the shoulder/upper arm in a contralateral fashion.
  Interventions: Drug: Testosterone gel (FE 999303)

INTERVENTIONS:
Drug: Testosterone gel (FE 999303)

SUMMARY:
This is a Phase 3 clinical trial in adult hypogonadal males with baseline serum testosterone concentrations <300 ng/dL. The purpose of this study is to evaluate the safety and efficacy of testosterone gel (2%) delivered using an applicator.

ELIGIBILITY:
Inclusion Criteria:

1. Males between 18-75 years of age
2. Two screening serum testosterone values less than 300 ng/dL
3. One or more symptoms of testosterone deficiency

Exclusion Criteria:

1. Previous use of the investigational product
2. Use of any investigational product within 30 days prior to screening and during the study
3. BMI less than 18 kg/m^2 or more than 35 kg/m^2
4. Prostatic mass(es)
5. Generalized skin irritation or skin disease
6. Lower urinary tract obstruction
7. Myocardial infarction or cerebrovascular accident in the last 6 months
8. Unstable angina or congestive heart failure
9. Thromboembolic disorders
10. Sleep apnea
11. Hyperparathyroidism or uncontrolled diabetes
12. Untreated moderate to severe depression
13. History of testicular, prostate, or breast cancer
14. HIV, Hepatitis B, or Hepatitis C positive
15. PSA more or equal to 3 ng/mL
16. Use of any medications that could be considered anabolic
17. Use of estrogens, Gonadotropin Releasing Hormone agonists/antagonists, antiandrogens, or human Growth Hormone
18. Chronic use of any drug of abuse
19. Involvement in a sport in which there is a screening for anabolic steroids
20. Not willing to use adequate contraception during the study
21. Partner is pregnant and/or breast feeding
22. Partner has a history of breast, uterine or ovarian cancer

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (19):
- United States (17):
  - Medical Affiliated Research Cente, Huntsville, Alabama
  - California Professional Research, Newport Beach, California
  - San Diego Sexual Medicine, San Diego, California
  - Connecticut Clinical Research, Middlebury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Michigan Institute of Urology, Saint Clair Shores, Michigan
  - Quality Clinical Research, Omaha, Nebraska
  - Premier Urology Associates, Lawrenceville, New Jersey
  - University Urology, New York, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - PMG Research of Wilmington, Winston-Salem, North Carolina
  - Tristate Urologic Services, Cincinnati, Ohio
  - Omega Medical Research, Warwick, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Clinical Research Associates, Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
- Canada (2):
  - St. Joseph's Healthcare, London, Ontario
  - Private Practice and Clinical Research, North Bay, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 19 study centers (17 in the US and 2 in Canada).
Pre-assignment Details: Of the 656 screened subjects, 180 subjects were enrolled into the study.
Period: Overall Study
Arm/Group | Testosterone Gel (FE 999303)
Started | 180
Completed | 172
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Consent Withdrawn | 1
Not completed — Investigator/Sponsor decision | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 2
Not completed — Participant Left for More Than 3 Months | 1
Not completed — Could Not Continue Due to Time Constrain | 1

BASELINE CHARACTERISTICS:
Population: Demographics analysis was done on the intent-to-treat (ITT) population consisting of all participants who received at least one dose of investigational medicinal product (IMP).
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 145
  >=65 years | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 164
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 157
  More than one race | 0
  Unknown or Not Reported | 1
Height, Continuous [Mean (Standard Deviation); unit: Inches] | 70.3 (2.8)
Weight, Continuous [Mean (Standard Deviation); unit: pounds] | 211.3 (30.1)
BMI, Continuous [Mean (Standard Deviation); unit: kg/m^2] | 30 (3.4)
Total International Index of Erectile Function (IIEF) Score [Mean (Standard Deviation); unit: units on a scale] — IIEF questionnaire have 15 questions (Q) divided into 5 domains-
  1. Erectile function (6 items, Q 1-5 and 15) (Score range: 1-30)
  2. Orgasmic function (2 items, Q 9-10) (Score range: 0-10)
  3. Sexual desire (2 items, Q 11-12) (Score range: 2-10)
  4. Intercourse satisfaction (3 items, Q 6-8) (Score range: 0-15)
  5. Overall satisfaction (2 items, Q 13-14) (Score range: 2-10)
  Total score was calculated by summing up scores of each domain and ranged from 5-75. Low score indicates severe dysfunction and a high score indicates no dysfunction in sexual function.
  units on a scale | 31.9 (18.4)
Multidimensional Assessment of Fatigue [Mean (Standard Deviation); unit: units on a scale] — The MAF have 16 questions (Q) divided into 4 domains:
  1. Severity (Q 1-2) (Score range [SR]: 2-20)
  2. Distress (Q 3) (SR: 1-10)
  3. Degree of interference in activities of daily living (Q 4-14) (SR: 11-110)
  4. Timing (Q 15-16) (SR: 5-20)
  First 14 Q are scored from 1-10. Questions 15-16 are scored from 1-4 and converted to 1-10 scale by multiplying each score by 2.5. Lower score in each domain indicates improvement in fatigue.
  GFI was calculated by summing up scores of Q 1, 2, 3, average of 4-14, and revised score of 15. Range of GFI: 1 (no fatigue) to 50 (severe fatigue).
  units on a scale
    Severity domain | 11.9 (5.5)
    Distress domain | 4.9 (2.8)
    Degree of interference domain | 48.9 (24.3)
    Timing domain | 12.8 (3.1)
    Global Fatigue Index (GFI) | 27.2 (12.6)
Short Form -12 (SF-12) Health survey [Mean (Standard Deviation); unit: units on a scale] — Data collected from the SF-12 questionnaire, based on the norm-based scores is used to assess improvement in the psychometrically-based physical component summary (PCS) and mental component summary (MCS). Both PCS and MCS contains four subdomains (A total of 12 questions).
  PCS and MCS composite scores are computed using the scores of the 12 questions and transforming these to range from 0-100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health. Positive change from baseline indicates improvement in physical and mental health.
  units on a scale
    Physical Component Summary | 47.5 (9.6)
    Mental Component Summary | 43.0 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects on Day 90 Whose Cavg (0-24) Serum Total Testosterone Levels Are Between 300 and 1050 ng/dL
Description: The data were presented using descriptive statistics. No statistical analysis was performed.
Time Frame: Day 90
Population: Full Analysis set (FAS) population was used which comprised of subjects who had any available pharmacokinetic (PK) data for testosterone on Day 90.
Measure: Number; unit: percentage of participants
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 172
percentage of participants
  23 mg | 2.9
  46 mg | 4.7
  69 mg | 77.9
  Overall | 85.5

2. Secondary Outcome: The Percentage of Participants on Day 1 Whose Serum Cavg (0-24) Serum Total Testosterone Levels Are Between 300 and 1050 ng/dL
Description: The data were presented using descriptive statistics. No statistical analysis was performed.
Time Frame: Day 1
Population: FAS population was used which comprised of subjects who had any available PK data for testosterone on Day 90.
Measure: Number; unit: percentage of participants
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 172
percentage of participants | 51.7

3. Secondary Outcome: Pharmacokinetics of Total Testosterone Measuring Area Under the Concentration-time Curve From the Last Dose and 24 Hours Post-dose (AUCτ)
Description: A validated high pressure liquid chromatography with tandem mass spectrometry detection (LC/MS/MS) method was used to determine the levels of total testosterone.
Time Frame: Day 1; Day 90
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Mean (Standard Deviation); unit: ng*hr/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
ng*hr/dL
  Day 1; 46 mg (n=180) | 7,616 (2,242)
  Day 90; 23 mg (n=5) | 12,433 (3,100)
  Day 90; 46 mg (n=12) | 9,835 (3,831)
  Day 90; 69 mg (n=155) | 11,967 (4,439)
  Day 90; all doses (n=172) | 11,825 (4,382)

4. Secondary Outcome: Pharmacokinetics of Total Testosterone Measuring Time of Maximum Observed Concentration (Tmax)
Description: A validated LC/MS/MS method was used to determine the levels of total testosterone.
Time Frame: Day 1; Day 90
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Median (Full Range); unit: hour
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
hour
  Day 1; 46 mg (n=180) | 4 [0 to 24]
  Day 90; 23 mg (n=5) | 4 [1.75 to 18]
  Day 90; 46 mg (n=12) | 2.01 [0 to 8]
  Day 90; 69 mg (n=155) | 2.03 [0 to 17.5]
  Day 90; all doses (n=172) | 2.03 [0 to 18]

5. Secondary Outcome: Pharmacokinetics of Total Testosterone Measuring Maximum Concentration Observed (Cmax)
Description: A validated LC/MS/MS method was used to determine the levels of total testosterone.
Time Frame: Day 1; Day 90
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
ng/dL
  Day 1; 46 mg (n=180) | 490 (234)
  Day 90; 23 mg (n=5) | 944 (253)
  Day 90; 46 mg (n=12) | 916 (514)
  Day 90; 69 mg (n=155) | 1,432 (1,050)
  Day 90; all doses (n=172) | 1,382 (1,017)

6. Secondary Outcome: Pharmacokinetics of Total Testosterone Measuring Average Steady State Concentration (Cave)
Description: A validated LC/MS/MS method was used to determine the levels of total testosterone.
Time Frame: Day 1; Day 90
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
ng/dL
  Day 1; 46 mg (n=180) | 316 (92)
  Day 90; 23 mg (n=5) | 515 (132)
  Day 90; 46 mg (n=12) | 407 (160)
  Day 90; 69 mg (n=155) | 495 (184)
  Day 90; all doses (n=172) | 489 (182)

7. Secondary Outcome: Pharmacokinetics of Total Testosterone Measuring Minimum Concentration Observed (Cmin)
Description: A validated LC/MS/MS method was used to determine the levels of total testosterone.
Time Frame: Day 1; Day 90
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
ng/dL
  Day 1; 46 mg (n=180) | 201 (65)
  Day 90; 23 mg (n=5) | 317 (112)
  Day 90; 46 mg (n=12) | 219 (76)
  Day 90; 69 mg (n=155) | 222 (89)
  Day 90; all doses (n=172) | 225 (90)

8. Secondary Outcome: Pharmacokinetics of Total Testosterone Measuring Time of Minimum Observed Concentration (Tmin)
Description: A validated LC/MS/MS method was used to determine the levels of total testosterone.
Time Frame: Day 1; Day 90
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Median (Full Range); unit: hour
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
hour
  Day 1; 46 mg (n=180) | 0 [0 to 24.0]
  Day 90; 23 mg (n=5) | 8.00 [0 to 18.0]
  Day 90; 46 mg (n=12) | 12.1 [0 to 24.0]
  Day 90; 69 mg (n=155) | 12.0 [0 to 24.0]
  Day 90; all doses (n=172) | 12.0 [0 to 24.0]

9. Secondary Outcome: Pharmacokinetics of DHT (Dihydrotestosterone) Measuring AUCτ
Description: A validated LC/MS/MS method was used to determine the levels of DHT.
Time Frame: Day 1; Day 90
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Mean (Standard Deviation); unit: ng*hr/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
ng*hr/dL
  Day 1; 46 mg (n=180) | 982 (588)
  Day 90; 23 mg (n=5) | 1,537 (263)
  Day 90; 46 mg (n=12) | 1,329 (593)
  Day 90; 69 mg (n=155) | 1,604 (698)
  Day 90; all doses (n=172) | 1,582 (683)

10. Secondary Outcome: Pharmacokinetics of DHT Measuring Tmax
Description: A validated LC/MS/MS method was used to determine the levels of DHT.
Time Frame: Day 1; Day 90
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Median (Full Range); unit: hour
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
hour
  Day 1; 46 mg (n=180) | 6 [0 to 24]
  Day 90; 23 mg (n=5) | 4.08 [2 to 18]
  Day 90; 46 mg (n=12) | 2.11 [0 to 8]
  Day 90; 69 mg (n=155) | 3.98 [0 to 24]
  Day 90; all doses (n=172) | 3.97 [0 to 24]

11. Secondary Outcome: Pharmacokinetics of DHT Measuring Cmax
Description: A validated LC/MS/MS method was used to determine the levels of DHT.
Time Frame: Day 1; Day 90
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
ng/dL
  Day 1; 46 mg (n=180) | 58.7 (40.1)
  Day 90; 23 mg (n=5) | 92.1 (21.9)
  Day 90; 46 mg (n=12) | 82.5 (37.7)
  Day 90; 69 mg (n=155) | 108 (51.0)
  Day 90; all doses (n=172) | 106 (50)

12. Secondary Outcome: Pharmacokinetics of DHT Measuring Cave
Description: A validated LC/MS/MS method was used to determine the levels of DHT.
Time Frame: Day 1; Day 90
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
ng/dL
  Day 1; 46 mg (n=180) | 40.8 (24.5)
  Day 90; 23 mg (n=5) | 63.7 (11.3)
  Day 90; 46 mg (n=12) | 55.1 (24.7)
  Day 90; 69 mg (n=155) | 66.3 (29.0)
  Day 90; all doses (n=172) | 65.4 (28.4)

13. Secondary Outcome: Pharmacokinetics of DHT Measuring Cmin
Description: A validated LC/MS/MS method was used to determine the levels of DHT.
Time Frame: Day 1; Day 90
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
ng/dL
  Day 1; 46 mg (n=180) | 18.0 (9.9)
  Day 90; 23 mg (n=5) | 45.4 (10.8)
  Day 90; 46 mg (n=12) | 35.7 (14.0)
  Day 90; 69 mg (n=155) | 42.8 (22.0)
  Day 90; all doses (n=172) | 42.4 (21.3)

14. Secondary Outcome: Pharmacokinetics of DHT Measuring Tmin
Description: A validated LC/MS/MS method was used to determine the levels of DHT.
Time Frame: Day 1; Day 90
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Median (Full Range); unit: hour
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
hour
  Day 1; 46 mg (n=180) | 0 [0 to 24.0]
  Day 90; 23 mg (n=5) | 8.00 [0 to 18.0]
  Day 90; 46 mg (n=12) | 16.0 [0 to 24.0]
  Day 90; 69 mg (n=155) | 12.0 [0 to 24.0]
  Day 90; all doses (n=172) | 12.0 [0 to 24.0]

15. Secondary Outcome: Change From Baseline in the International Index of Erectile Dysfunction (IIEF) Questionnaire
Description: Data collected from the five domains of sexual functions were summarized by descriptive statistics. The domains are:
  1. Erectile function (6 items, questions 1-5 and 15) (Score range: 1-30)
  2. Orgasmic function (2 items, questions 9-10) (Score range: 0-10)
  3. Sexual desire (2 items, questions 11-12) (Score range: 2-10)
  4. Intercourse satisfaction (3 items, questions 6-8) (Score range: 0-15)
  5. Overall satisfaction (2 items, questions 13-14) (Score range: 2-10)
  A score of 0-5 is awarded to questions 1 to 10 and a score of 1-5 is awarded to questions 11 to 15. Total score was calculated by summing up scores of each domain and ranged from 5 to 75. Low score indicates severe dysfunction and a high score indicates no dysfunction in sexual function.
Time Frame: Day 91
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
units on a scale | 13.8 (17.1)

16. Secondary Outcome: Change From Baseline in the Multidimensional Assessment of Fatigue (MAF) Questionnaire
Description: The MAF contains four sub-domains:
  1. Severity (2 items, questions 1-2) (Score range: 2-20)
  2. Distress (1 item, question 3) (Score range: 1-10)
  3. Degree of interference in activities of daily living (11 items, questions 4-14) (Score range: 11-110)
  4. Timing (2 items, questions 15-16) (Score range: 5-20)
  A score of 1-10 is awarded to each of the 14 questions across the 3 domains. The timing domain is categorical and was converted to 1-10 scale by multiplying each score by 2.5. Lower score in each domain indicates improvement in fatigue.
  To calculate GFI : Score of question 15 is converted to a 0-10 scale by multiplying each score by 2.5 and then sum questions 1, 2, 3, average of 4-14, and newly scored question 15. A score of zero is assigned to question 2-16, if patient select 'no fatigue' to question 1. Question 16 is not included in GFI calculation. Range of GFI: 1 (no fatigue) to 50 (severe fatigue).
  The data were presented using descriptive statistics.
Time Frame: Day 91
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
units on a scale
  Severity domain score | -5.3 (5.3)
  Distress domain score | -2.0 (2.7)
  Degree of interference domain score | -18.9 (22.0)
  Timing domain score | -2.8 (3.5)
  GFI score | -11.4 (11.9)

17. Secondary Outcome: Change From Baseline in the SF-12 Health Questionnaire
Description: Data collected from the SF-12 questionnaire was used to assess improvement in the psychometrically-based physical component summary (PCS) and mental component summary (MCS). Both PCS and MCS contains four sub-domains:
  PCS: General Health (1 item), Physical Functioning (2 items), Role-Physical (2 items), Bodily Pain (1 item)
  MCS: Role-Emotional (2 items), Mental Health (2 items), Vitality (1 item), Social Functioning (1 item)
  The scale scores are calculated by summing responses across scale items and then transforming these raw scores to a 0-100 scale. Computerized scoring algorithms are used to produce norm-based scores for each scale (mean of 50 and standard deviation of 10) as well as the PCS and MCS summary scores. A zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
  The data were presented using descriptive statistics.
Time Frame: Day 91
Population: ITT population was used which comprised of all participants who received at least one dose of IMP.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 180
units on a scale
  Physical Component Summary (PCS) | 3.7 (7.1)
  Mental Component Summary (MCS) | 7.9 (10.4)

ADVERSE EVENTS:
Time Frame: Overall study period (From Day -45 [screening] to Day 91 [last visit])
Description: The treatment-emergent adverse event, defined as any adverse event occurring after start of IMP administration and within the time of residual drug effect (5 days), or a pre-treatment adverse event or pre-existing medical condition that worsens in intensity after start of IMP and within the time of residual drug effect, were presented.
Arm/Group | Testosterone Gel (FE 999303)
Serious Adverse Events (participants affected / at risk) | 3/180
Other Adverse Events (participants affected / at risk) | 62/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Gel (FE 999303) (N=180)
Myocardial infarction (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Compression fracture lumbar spine (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone Gel (FE 999303) (N=180)
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Inflammation (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Periumbilical abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Muscle injury (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 2
Haematocrit increased (Investigations) | 1
Haemoglobin increased (Investigations) | 2
Heart rate irregular (Investigations) | 1
Prostatic specific antigen increased (Investigations) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Calculus bladder (Renal and urinary disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Ejaculation failure (Reproductive system and breast disorders) | 1
Epididymitis (Reproductive system and breast disorders) | 1
Scrotal cyst (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 2
Cataract operation (Surgical and medical procedures) | 1
Dental operation (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 3
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.